CLINICAL TRIAL: NCT04688489
Title: Randomized Controlled Trial on the Effect of Carbloading and Maltodextrin on the Level of Function in Patients With Apoplexia
Brief Title: Effect of Carbloading and Maltodextrin on the Level of Function in Patients With Apoplexia
Acronym: ApoCarb
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Jens Rikardt Andersen, Associate Professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H-20018258
Record Dates: First submitted 2020-11-17; First posted 2020-12-30 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Apoplexy; Brain
Keywords: carbohydrates; rehabilitation; high-carbohydrate diet
MeSH Terms: conditions — Stroke | interventions — maltodextrin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): The intervention consists of a supplement of maltodextrin at training episodes combined with added dietary carbohydrates at all meals
  Interventions: Dietary Supplement: Carbloading and maltodextrin
- Control (No Intervention): The control receives no intervention. Standard treatment will be administered.

INTERVENTIONS:
Dietary Supplement: Carbloading and maltodextrin — The intervention is a dietary intervention that consists of a supplement of maltodextrin and added dietary carbohydrates. The supplement (20 g for women and 30 g for men) will be given to patients before and after a scheduled training, while the carbohydrates are given with meals. The extra carbohydrates given at meal time consists of extra potatoes, rice, bread, fruit, juice or other carbohydrate-rich food items.
  Arms: Intervention

SUMMARY:
The study will investigate the potential effect of a supplement of maltodextrin and added dietary carbohydrates on the level of function in patients with apoplexia. The study has an intervention group and a control group. The study is randomized, but not blinded. The primary outcome is level of function measured with Barthel-100. Besides the primary outcome there are several secondary outcomes (see detailed description). All patients are recruited from Rigshospitalet, Glostrup.

DETAILED DESCRIPTION:
The study will investigate the potential effect of a supplement of maltodextrin (20 g for women and 30 g for men) and added dietary carbohydrates on the level of function in patients with apoplexia. The study has an intervention group and a control group. The study is randomized, but not blinded. The primary outcome is level of function measured with Barthel-100. Secondary outcomes are: training intensity, duration and frequency; length of stay; self-training (training without a therapist) and patient's experienced fatigue; and patient's experienced pain. All patients are recruited from Rigshospitalet, Glostrup. The supplement will be administered before and after each training session with a therapist. The supplement is a powder desolved in a glass of juice. The nursing staff will add extra carbohydrates to the patient's meals in the form of potatoes, rice, bread, fruit or other carbohydrate rich food items. All meals will be noted daily and validated the following day by the primary investigators.

ELIGIBILITY:
Inclusion Criteria:

* Patients with apoplexia who are declared suited for rehabilitation at Afs. Neurologisk Afdeling N 35 - Apopleksi or Afs. Neurologisk Afdeling N 45 - Apopleksi, Rigshospitalet, Glostrup
* Patient must be able to consent participation
* Age 50+ years
* Must be able to understand danish
* Must be relevant for physio- or occupational therapy

Exclusion Criteria:

* Diabetes Mellitus type I og type II
* Enteral nutrition (tube feeding)
* Barthel-100 over 80 points

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Difference between inclusion and discharge in score | 8 weeks
  Measured with Barthel100 by the nursing staff

SECONDARY OUTCOMES:
Length of stay (days) | 8 weeks
  Measured in full days
Intensity of training (score) | 8 weeks
  Assessed by the therapists who trained with the patient.
Duration of training (hours) | 8 weeks
  Assessed by the therapists after every training. Noted i the same document as "intensity of training"
Frequency of training with therapist (episodes/week) | 8 weeks
  Assessed by the therapists after every training.
Level of experienced fatique (VAS - score) | 8 weeks
  Measured by a VAS-fatigue scale.
Level of experienced post-work out muscle soreness (VAS - score) | 8 weeks
  Measured by a VAS-pain scale.
Level of physical activity during hospital admission - daily score | 8 weeks
  Noted on a document by the patient or the study officials.

CONTACTS AND LOCATIONS:
Overall Officials: Helle Klingenberg Iversen, Principal Investigator — Neurologisk Klinik, Rigshospitalet Glostrup
Locations (1):
- Rigshospitalet, Glostrup, Glostrup, Region Sjælland, Denmark

IPD SHARING:
Plan to Share IPD: No